CLINICAL TRIAL: NCT02387580
Title: A Phase I Bioavailability Study of Selected Oral Prototype Granule Formulations of OZ439 in Healthy Subjects, to Evaluate the Pharmacokinetics of OZ439 When Co-Administered With Piperaquine Phosphate Tablets in the Fasted State
Brief Title: Bioavailability Study of Oral OZ439 Prototype Granule Formulations Administered With Piperaquine Phosphate (PQP) Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMV_OZ439_15_001
Record Dates: First submitted 2015-03-05; First posted 2015-03-13 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Malaria
Keywords: Malaria; Bioavailability; Formulation
MeSH Terms: conditions — Malaria | interventions — artefenomel; tocophersolan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Regimen A: OZ439 + TPGS and PQP (Active Comparator): 800 mg OZ439 + TPGS granules (oral suspension 240 mL volume and 100 mL rinse volume) and 960 mg (3 × 320 mg) PQP tablets
  Interventions: Drug: OZ439 + TPGS; Drug: PQP
- Regimen B: OZ439 Prototype 1 and PQP - 110mL (Experimental): 800 mg OZ439 Prototype 1 granules (oral suspension 60 mL volume and 50 mL rinse volume) and 960 mg (3 × 320 mg) PQP tablets
  Interventions: Drug: OZ439 Prototype 1; Drug: PQP
- Regimen C: OZ439 Prototype 3 and PQP - 110mL (Experimental): 800 mg OZ439 Prototype 3 granules (oral suspension 60 mL volume and 50 mL rinse volume) and 960 mg (3 × 320 mg) PQP tablets
  Interventions: Drug: OZ439 Prototype 3; Drug: PQP
- Regimen D: OZ439 + TPGS and PQP (Active Comparator): 800 mg OZ439 + TPGS granules (oral suspension 240 mL volume and 100 mL rinse volume) and 960 mg (3 × 320 mg) PQP tablets
  Interventions: Drug: OZ439 + TPGS; Drug: PQP
- Regimen E: OZ439 Prototype 1 or 3 and PQP - XmL (Experimental): 800 mg OZ439 Prototype 1 or 3 granules (oral suspension and rinse volume to be determined) and 960 mg (3 × 320 mg) PQP tablets
  Interventions: Drug: OZ439 Prototype 1; Drug: PQP
- Regimen F: OZ439 Prototype 1 or 3 and PQP - XmL (Experimental): 800 mg OZ439 Prototype 1 or 3 granules (oral suspension and rinse volume to be determined) and 960 mg (3 × 320 mg) PQP tablets
  Interventions: Drug: OZ439 Prototype 3; Drug: PQP

INTERVENTIONS:
Drug: OZ439 + TPGS
  Other Names: 800 mg OZ439 + TPGS Reference Treatment
  Arms: Regimen A: OZ439 + TPGS and PQP; Regimen D: OZ439 + TPGS and PQP
Drug: OZ439 Prototype 1
  Other Names: OZ439 Granules Prototype 1 Granules Formulation
  Arms: Regimen B: OZ439 Prototype 1 and PQP - 110mL; Regimen E: OZ439 Prototype 1 or 3 and PQP - XmL
Drug: OZ439 Prototype 3
  Other Names: OZ439 Granules Prototype 3 Granules Formulation
  Arms: Regimen C: OZ439 Prototype 3 and PQP - 110mL; Regimen F: OZ439 Prototype 1 or 3 and PQP - XmL
Drug: PQP
  Other Names: PQP 960 mg tablets

SUMMARY:
This is a single-centre, 2-part, randomised, single-dose parallel group study in healthy male subjects and female subjects of non-childbearing potential.

DETAILED DESCRIPTION:
Parts 1 and 2 will be randomised with 8 subjects receiving each regimen:

Part 1:

* Regimen A: Reference: 800 mg OZ439 + α-Tocopherol polyethylene glycol 1000 succinate (TPGS) granules (oral suspension 240 mL volume and 100 mL rinse volume) and 960 mg (3 × 320 mg) PQP tablets
* Regimen B: Prototype 1: 800 mg OZ439 granules (oral suspension 60 mL volume and 50 mL rinse volume) and 960 mg (3 × 320 mg) PQP tablets
* Regimen C: Prototype 3: 800 mg OZ439 granules (oral suspension 60 mL volume and 50 mL rinse volume) and 960 mg (3 × 320 mg) PQP tablets

There will be an interim decision after Part 1 to determine the formulation prototypes and the oral suspension volume to be administered in Part 2.

Part 2

* Regimen D: Reference: 800 mg OZ439 + TPGS granules (oral suspension 240 mL volume and 100 mL rinse volume) and 960 mg (3 × 320 mg) PQP tablets
* Regimen E: Prototype 1 or 3: 800 mg OZ439 granules (oral suspension and rinse volume to be determined) and 960 mg (3 × 320 mg) PQP tablets
* Regimen F: Prototype 1 or 3: 800 mg OZ439 granules (oral suspension and rinse volume to be determined) and 960 mg (3 × 320 mg) PQP tablets

ELIGIBILITY:
Inclusion Criteria:

* Healthy males, or healthy females of non-childbearing potential ie surgically sterilised or post-menopausal
* Body mass index of 18.0 to 30.0 kg/m2 inclusive. Total body weight >50 kg at screening.
* Must agree to use an adequate method of contraception.
* Normal laboratory tests as judged by the Investigator.
* Must have QTcF ≤450 ms, QTcB ≤450 ms for male subjects, QTcF ≤470 ms, QTcB ≤470 ms for female subjects and PR interval ≤200 ms for screening and pre-dose ECG measurements.

Exclusion Criteria:

* Male subjects who have currently pregnant partners or who have partners planning to be pregnant.
* Evidence or history of clinically significant disease, or current infection.3.
* Clinically relevant abnormalities in the ECG.
* Family history of sudden death or of congenital prolongation of the QTc interval or known congenital prolongation of the QTc interval or any clinical condition known to prolong the QTc interval.
* History of symptomatic cardiac arrhythmias or with clinically relevant bradycardia, heart rate ≤39 bpm.
* Electrolyte disturbances, particularly hypokalaemia, hypocalcaemia or hypomagnesaemia.
* History of any drug or alcohol abuse in the past 2 years prior to screening.
* Receipt of an investigational drug or participation in another clinical research study within 90 days prior to drug administration.
* Use of any prescription or non-prescription medications, vitamins, herbal supplements or dietary supplements, including protein supplements, within 14 days prior to the first dose of study drug.
* Positive hepatitis B surface antigen, hepatitis C virus antibody or human immunodeficiency virus results.
* Clinically significant abnormal biochemistry, haematology or urinalysis.
* Positive urine drug screen result.
* History of intolerance or hypersensitivity to PQP or any 4-aminoquinoline, or ascertained or presumptive hypersensitivity to the active principle and/or formulation ingredients; history of anaphylaxis to drugs or allergic reactions in general, that the investigator considers may affect the outcome of the study.
* Presence or history of allergy requiring treatment; hayfever is allowed unless it is active.
* Donation or loss of >400 mL of blood within 90 days prior to drug administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Macintyre, PhD, Study Director — Medicines for Malaria Ventire
Locations (1):
- Quotient Clinical, Nottingham, Nottinghamshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Regimen E: OZ439 Prototype 1 or 3 and PQP - 220mL; Regimen F: OZ439 Prototype 1 or 3 and PQP - 220mL: 800 mg OZ439 Prototype 1 or 3 granules (120mL oral suspension and 100mL rinse volume) and 960 mg (3 × 320 mg) PQP tablets
Period: Overall Study
Arm/Group | Regimen A: OZ439 + TPGS and PQP | Regimen B: OZ439 Prototype 1 and PQP - 110mL | Regimen C: OZ439 Prototype 3 and PQP - 110mL | Regimen D: OZ439 + TPGS and PQP | Regimen E: OZ439 Prototype 1 or 3 and PQP - 220mL | Regimen F: OZ439 Prototype 1 or 3 and PQP - 220mL
Started | 8 | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 7 | 8 | 8
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population was to include all subjects who received at least 1 dose of IMP. All 48 subjects met the criteria for inclusion in the safety population
Groups:
- Regimen E: OZ439 Prototype 1 or 3 and PQP - 220mL: 800 mg OZ439 Prototype 1 or 3 granules (120 mL oral suspension and 100 mL rinse volume) and 960 mg (3 × 320 mg) PQP tablets
- Regimen F: OZ439 Prototype 1 or 3 and PQP - 220mL: 800 mg OZ439 Prototype 1 or 3 granules (120 mL oral suspension and 100 mL rinse volume ) and 960 mg (3 × 320 mg) PQP tablets
- Total: Total of all reporting groups
Arm/Group | Regimen A: OZ439 + TPGS and PQP | Regimen B: OZ439 Prototype 1 and PQP - 110mL | Regimen C: OZ439 Prototype 3 and PQP - 110mL | Regimen D: OZ439 + TPGS and PQP | Regimen E: OZ439 Prototype 1 or 3 and PQP - 220mL | Regimen F: OZ439 Prototype 1 or 3 and PQP - 220mL | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (8.9) | 34.5 (12.7) | 34.9 (9.8) | 32.0 (12.9) | 31.3 (12.9) | 30.1 (7.0) | 32.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Male | 8 | 8 | 8 | 8 | 7 | 8 | 47
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8 | 8 | 8 | 8 | 8 | 8 | 48

OUTCOME MEASURES:

1. Primary Outcome: OZ439 Cmax
Description: OZ439 Maximum observed concentration
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72, 96 and 168 hours post-dose
Population: The PK population was to include all valid profiles from subjects dosed with IMP. 45 subjects were included in the PK population. 3 subjects vomited approximately 1 to 2 h after dosing and were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Regimen A: OZ439 + TPGS and PQP | Regimen B: OZ439 Prototype 1 and PQP - 110mL | Regimen C: OZ439 Prototype 3 and PQP - 110mL | Regimen D: OZ439 + TPGS and PQP | Regimen E: OZ439 Prototype 1 or 3 and PQP - 220mL | Regimen F: OZ439 Prototype 1 or 3 and PQP - 220mL
Number analyzed (Participants) | 7 | 8 | 8 | 6 | 8 | 8
ng/mL | 1600 (36.6) | 824 (38.3) | 616 (49.4) | 1530 (13.2) | 999 (40.8) | 730 (35.7)

2. Primary Outcome: OZ439 AUC(0-168 h)
Description: OZ439 Area under the plasma concentration (AUC) versus time curve
Time Frame: pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72, 96 and 168 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Regimen A: OZ439 + TPGS and PQP | Regimen B: OZ439 Prototype 1 and PQP - 110mL | Regimen C: OZ439 Prototype 3 and PQP - 110mL | Regimen D: OZ439 + TPGS and PQP | Regimen E: OZ439 Prototype 1 or 3 and PQP - 220mL | Regimen F: OZ439 Prototype 1 or 3 and PQP - 220mL
Number analyzed (Participants) | 7 | 8 | 8 | 6 | 8 | 8
ng*h/mL | 15300 (26.1) | 7920 (26.4) | 5610 (38.1) | 14000 (29.6) | 9550 (57.5) | 7100 (45.7)

3. Primary Outcome: Piperaquine Cmax
Description: Piperaquine Maximum observed concentration
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72, 96 and 168 hours and Day36 post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Regimen A: OZ439 + TPGS and PQP | Regimen B: OZ439 Prototype 1 and PQP - 110mL | Regimen C: OZ439 Prototype 3 and PQP - 110mL | Regimen D: OZ439 + TPGS and PQP | Regimen E: OZ439 Prototype 1 or 3 and PQP - 220mL | Regimen F: OZ439 Prototype 1 or 3 and PQP - 220mL
Number analyzed (Participants) | 7 | 8 | 8 | 6 | 8 | 8
ng/mL | 183 (124.9) | 62.1 (154.4) | 100 (80.7) | 119 (52.1) | 91.8 (108.2) | 95.7 (81.5)

4. Primary Outcome: Piperaquine AUC(0-168 h)
Description: PQP Area under the plasma concentration versus time curve
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72, 96 and 168 hours and Day36 post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Regimen A: OZ439 + TPGS and PQP | Regimen B: OZ439 Prototype 1 and PQP - 110mL | Regimen C: OZ439 Prototype 3 and PQP - 110mL | Regimen D: OZ439 + TPGS and PQP | Regimen E: OZ439 Prototype 1 or 3 and PQP - 220mL | Regimen F: OZ439 Prototype 1 or 3 and PQP - 220mL
Number analyzed (Participants) | 7 | 8 | 8 | 6 | 8 | 8
ng*h/mL | 3740 (61.2) | 1940 (69.5) | 2980 (47.6) | 2860 (40.2) | 2550 (47.8) | 2470 (60.8)

ADVERSE EVENTS:
Time Frame: Up to Day 36 post-dose.
Description: The safety population was to include all subjects who received at least 1 dose of IMP.
  All 48 subjects met the criteria for inclusion in the safety population.
Arm/Group | Regimen A: OZ439 + TPGS and PQP | Regimen B: OZ439 Prototype 1 and PQP - 110mL | Regimen C: OZ439 Prototype 3 and PQP - 110mL | Regimen D: OZ439 + TPGS and PQP | Regimen E: OZ439 Prototype 1 or 3 and PQP - 220mL | Regimen F: OZ439 Prototype 1 or 3 and PQP - 220mL
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 4/8 | 3/8 | 6/8 | 5/8 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A: OZ439 + TPGS and PQP (N=8) | Regimen B: OZ439 Prototype 1 and PQP - 110mL (N=8) | Regimen C: OZ439 Prototype 3 and PQP - 110mL (N=8) | Regimen D: OZ439 + TPGS and PQP (N=8) | Regimen E: OZ439 Prototype 1 or 3 and PQP - 220mL (N=8) | Regimen F: OZ439 Prototype 1 or 3 and PQP - 220mL (N=8)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Investigator considered the SAE to be unrelated to IMP due to intake of other pharmacological agents known to induce atrial fibrillation ie Beechams all-in-one and possibly cocaine.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A: OZ439 + TPGS and PQP (N=8) | Regimen B: OZ439 Prototype 1 and PQP - 110mL (N=8) | Regimen C: OZ439 Prototype 3 and PQP - 110mL (N=8) | Regimen D: OZ439 + TPGS and PQP (N=8) | Regimen E: OZ439 Prototype 1 or 3 and PQP - 220mL (N=8) | Regimen F: OZ439 Prototype 1 or 3 and PQP - 220mL (N=8)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epigastric Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary Hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal Allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Influenza Like Illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Quotient shall have the right to publish the results of the research, subject to the sponsor's prior written consent, which shall not be unreasonably withheld or delayed. Following the receipt of such consent, Quotient shall submit a copy of the proposed publication to the sponsor who shall have 30 days in which to request amendments thereto which, to the extent that such proposed amendments are reasonable, Quotient shall be obliged to incorporate prior to such publication.